CLINICAL TRIAL: NCT00799890
Title: Monocentric, Prospective, Doubleblind, Randomised/Stratified, Placebocontrolled Two-arm Study to Evaluate the Effect of Sunphenon EGCg (Main Component Epigallocatechin-Gallat) on the Increase of Brain Atrophy in the Cerebral Magnetic Resonance Tomography in a 36-months Treatment Time in Patients With Primary or Secondary Chronic-progressive Multiple Sclerosis
Brief Title: Sunphenon in Progressive Forms of Multiple Sclerosis
Acronym: SUPREMES
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Friedemann Paul (Other)
Collaborators: TAIYO EUROPE (Unknown)
Responsible Party: Sponsor-Investigator, Friedemann Paul, Prof. Dr., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUPREMES-01
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: primary or secondary chronic-progressive; sunphenon egcg; brain atrophy; T2 lesions
MeSH Terms: conditions — Multiple Sclerosis | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sunphenon (Experimental)
  Interventions: Drug: Sunphenon EGCG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sunphenon EGCG — 200-800mg (1-4 capsules)
  Other Names: Epigallo Catechin Gallate
  Arms: Sunphenon
Drug: Placebo — 1-4 capsules
  Arms: Placebo

SUMMARY:
The investigators hypothesize that an oral Sunphenon EGCg (Epigallocatechin-Gallat, EGCG) treatment is - due to its antiinflamatoric and neuroprotective potence - significantly more effective than an oral placebo treatment regarding following parameters: increase in brain atrophy, number of new T2-lesions in the cerebral magnetic resonance tomography, reduction of the NAA/Cr-ratio in MR-spectroscopy, progression of disability such as cognitive disorders in patients with MS.

DETAILED DESCRIPTION:
The hypotheses of our study are:

Sunphenon EGCg has an antiinflammatoric effect due to its impact on the T-cell-proliferation and the inhibition of the activity of NF-Kb.

Sunphenon EGCg has a neuroprotective effect due to its antioxidative potence as a radical scavenger.

A 30 month treatment with Sunphenon EGCg is safe and well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary chronic progressive multiple sclerosis (ms)
* EDSS 3-8
* Age 18-65

Exclusion Criteria:

* Relapsing-remitting ms
* Immunodulatoric or immunosuppressive therapy
* pretreatment with Mitoxantron, Natalizumab, Rituximab, Azathioprin <2 month before screening
* pretreatment with Glairameracetat or beta-Interferons <4 weeks before screening
* signs of hepatic dysfunction
* active ulcus ventriculi or duodeni
* neoplasias if not cured >1 year before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
brain atrophy | 36 months of treatment

SECONDARY OUTCOMES:
new T2 lesions | 36 months of treatment
reduction of the NAA/Cr-ratio in MR-spectroscopy | 36 months of treatment
progression of disability such as cognitive disorders | 36 months of treatment
number of AEs | 36 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Dr., Principal Investigator — Charite University (NeuroCure Clinical Research Center)
Locations (1):
- Charité Universitätsmedizin Berlin (NeuroCure Clinical Research Center), Berlin, Germany

REFERENCES:
- [Derived] Klumbies K, Rust R, Dorr J, Konietschke F, Paul F, Bellmann-Strobl J, Brandt AU, Zimmermann HG. Retinal Thickness Analysis in Progressive Multiple Sclerosis Patients Treated With Epigallocatechin Gallate: Optical Coherence Tomography Results From the SUPREMES Study. Front Neurol. 2021 Apr 28;12:615790. doi: 10.3389/fneur.2021.615790. eCollection 2021. PMID 33995239
- [Derived] Rust R, Chien C, Scheel M, Brandt AU, Dorr J, Wuerfel J, Klumbies K, Zimmermann H, Lorenz M, Wernecke KD, Bellmann-Strobl J, Paul F. Epigallocatechin Gallate in Progressive MS: A Randomized, Placebo-Controlled Trial. Neurol Neuroimmunol Neuroinflamm. 2021 Feb 23;8(3):e964. doi: 10.1212/NXI.0000000000000964. Print 2021 May. PMID 33622766
- See also: Related Info — http://www.charite.de/
- See also: Related Info — http://www.ncrc.de